CLINICAL TRIAL: NCT00594347
Title: Immunogenicity and Safety of a Booster Dose of Polysaccharide Pneumococcal Vaccine (Pneumo 23®) in 12 to 18 Months-Old Children Primed With Three Doses of Pneumococcal Conjugate Vaccine (Prevnar®) in Thailand.
Brief Title: Immunogenicity and Safety of a Booster Dose of Pneumo 23® in 12 to 18 Months-Old Children Primed With Prevnar
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PNA19
Record Dates: First submitted 2007-12-19; First posted 2008-01-15 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Streptococcus Pneumoniae
Keywords: Streptococcus pneumoniae
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Pneumo 23
  Interventions: Biological: Pneumo 23
- Group B (Active Comparator): Prevnar
  Interventions: Biological: Prevnar

INTERVENTIONS:
Biological: Pneumo 23 — Vaccine (Pneumo 23)
  Arms: Group A
Biological: Prevnar — Vaccine (Prevnar)
  Arms: Group B

SUMMARY:
The present study intends to investigate the use as a booster of a dose of sanofi pasteur's Pneumo 23 vaccine in the second year of life following 3-dose priming with Wyeth's Prevnar vaccine. The researchers will use a cohort of subjects who have received 3 doses of Prevnar® at 2, 4, 6 months of age in the context of the clinical study A3L12 on Hexavalent combined vaccine (DTaP-IPV-HB-PRP~T)

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to 18 months on the day of inclusion
* Informed consent form signed by the parent/legally acceptable representative and by an independent witness if requested by local Ethics Committee regulation or/and if the parent/legally acceptable representative is illiterate
* Child having completed the three-dose primary vaccination of Prevnar® in the hexavalent combined vaccine study (study A3L12).
* Subjects and parent/guardian able to attend all scheduled visits and comply with all study procedures

Exclusion Criteria:

* Participation in another clinical study investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the study vaccination
* Planned participation in another clinical study during the present study period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the study vaccine or to a vaccine containing any of the same substances
* Chronic illness at a stage that could interfere with study conduct or completion, in the opinion of the investigator
* Receipt of blood or blood-derived products since birth that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the study vaccination
* Planned receipt of any vaccine in the 4 weeks preceding or following study vaccination
* History of seizures Known personal Human Immunodeficiency Virus (HIV), Hepatitis B (HB) antigen or Hepatitis C seropositivity
* History of pneumococcal infection (confirmed either clinically, serologically or microbiologically)
* Previous booster vaccination against the pneumococcal disease with either the study vaccine(s) or another vaccine
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating IM vaccination
* Febrile illness (temperature ≥ 38°C) or moderate or severe acute illness/infection on the day of vaccination, according to investigator judgment.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 339 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety after booster administration of 23-valent polysaccharidic pneumococcal vaccine | 30 days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Thailand (2):
  - Bangkok
  - KhonKaen

REFERENCES:
- [Result] Thisyakorn U, Chokephaibulkit K, Kosalaraksa P, Benjaponpitak S, Pancharoen C, Chuenkitmongkol S. Immunogenicity and safety of 23-valent pneumococcal polysaccharide vaccine as a booster dose in 12- to 18-month-old children primed with 3 doses of 7-valent pneumococcal conjugate vaccine. Hum Vaccin Immunother. 2014;10(7):1859-65. doi: 10.4161/hv.28642. PMID 25424793
- See also: Related Info — http://www.sanofipasteur.com